CLINICAL TRIAL: NCT02061696
Title: A Randomized Controlled Trial to Assess Safety and Efficacy of AXERA 2 Access System Compared to Manual Compression
Brief Title: ARISTOCRAT-A Randomized Controlled Trial Evaluating Closure Following Access With the AXERA (Device Name) 2 Access System
Acronym: ARISTOCRAT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Device was modified and no longer available to investigator
Sponsor: Frank Saltiel (Other)
Collaborators: Borgess Medical Center (Unknown); Borgess Cardiology Group (Unknown); Borgess Heart Center for Excellence (Unknown)
Responsible Party: Sponsor-Investigator, Frank Saltiel, Borgess Heart Institute, Chairman, Borgess Research Institute
Organization: Borgess Research Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: BRI-001
Record Dates: First submitted 2014-01-30; First posted 2014-02-13 (Estimated); Results first posted 2017-08-18 (Actual); Last update posted 2018-05-23 (Actual); Status verified 2018-04

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Artery Disease; Coronary Disease; Heart disease; Cardiovascular Diseases; Arteriosclerosis; Atherosclerosis; Manual Compression
MeSH Terms: conditions — Coronary Artery Disease; Coronary Disease; Heart Diseases; Cardiovascular Diseases; Arteriosclerosis; Atherosclerosis | interventions — Vascular Access Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Manual Compression (Active Comparator): Standard manual compression at the access site applied as per standard of care protocol for sheath removal.
  Interventions: Procedure: Standard Manual Compression
- AXERA 2 Access System (Active Comparator): The Vascular Access device used is the AXERA 2 Access System for patients randomized to this arm.
  Interventions: Device: Vascular Access Device

INTERVENTIONS:
Device: Vascular Access Device — AXERA 2 Access System with Reduced Manual Compression
  Other Names: AXERA 2 Access System
  Arms: AXERA 2 Access System
Procedure: Standard Manual Compression — Closure procedure by Manual Compression
  Arms: Standard Manual Compression

SUMMARY:
The goal of the research study is to observe the clinical safety, effectiveness and patient satisfaction of the AXERA 2 Access System in subjects undergoing coronary angiographic and possible Percutaneous Coronary Intervention (PCI) through the femoral artery when compared to standard manual compression.

DETAILED DESCRIPTION:
The study is a single center 1:1 randomized controlled trial in subjects undergoing coronary angiography and PCI.

It is anticipated that the enrollment period for this study will be two years.

The post procedure follow up period is up to 37 days following the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Subject is between 18 and 85 years of age.
* Cardiac catheterization procedure is indicated with involving access through a 5 French (F) or 6 French (F) introducer in the femoral artery.
* Subject is able to ambulate without assistance prior to the procedure and can be expected to ambulate (20 feet) post-procedure.
* Subject or legally authorized representative has signed informed consent.

Exclusion Criteria:

* Subject is unable to routinely 20 feet without assistance (e.g. requires a walker or wheelchair to mobilize or has paralysis)
* Subject has an active systemic or cutaneous infection or inflammation (e.g. (septicemia at the time of the procedure).
* Subject undergoing emergent or urgent cardiac catheterization for acute myocardial infarction.
* Extensive calcification of the femoral artery as see on fluoroscopy.
* Subject has systemic hypertension unresponsive to treatment (>180mm Hg systolic and >110mm Hg diastolic).
* Subject has received thrombolytic therapy within the 72 hours prior to catheterization.
* Subject has known bleeding disorder,such as Factor 5 deficiency, Idiopathic thrombocytopenic purpura (ITP), thrombasthenia, Von Willebrand's disease.
* Is on warfarin with an International Ratio (INR)>1.5.
* Platelet count is < 100,000.
* Anemia (Hemoglobin <10 g/dl or Hematocrit<30%).
* Subject has compromised femoral artery access site.
* Subject procedure requires an introducer sheath size of > 6 French (F).
* Subject has had prior vascular surgery or vascular grafts at the femoral artery access site.
* Subject presents with hemodynamic instability or is in need of emergent surgery.
* Subject has received femoral artery closure on the target access vessel with a collagen/PEG closure device within 90 days.
* Subject has a pre-existing severe non-cardiac systemic disease or illness that results in an expected life expectancy of < 1 year.
* Subject is participating in an investigational drug or another device research study that interferes with the current research study endpoints.
* Pregnant or lactating subjects.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2014-01; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank Saltiel, MD, Principal Investigator — Chairman, Borgess Heart Institute
Locations (1):
- Borgess Medical Center, Kalamazoo, Michigan, United States

REFERENCES:
- [Background] Turi ZG, Wortham DC, Sampognaro GC, Kresock FD, Held JS, Smith RD, Veerina KK, Hinohara T, Kaki A. Use of a novel access technology for femoral artery catheterization: results of the RECITAL trial. J Invasive Cardiol. 2013 Jan;25(1):13-8. PMID 23293169

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Thirty-nine patients enrolled in the study.
Period: Overall Study
Arm/Group | Standard Manual Compression | AXERA 2 Access System
Started | 17 | 22
Completed | 17 | 22
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Manual Compression | AXERA 2 Access System | Total
Number analyzed (Participants) | 17 | 22 | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 13 | 23
  >=65 years | 7 | 9 | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 11 | 17 | 28
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 17 | 22 | 39

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Site-Related Major Adverse Events
Description: Observation of any major access site related complications (number of participants).
Time Frame: Up to 37 days post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Manual Compression | AXERA 2 Access System
Number analyzed (Participants) | 17 | 22
Participants | 0 | 0

2. Secondary Outcome: AXERA 2 Access System Success
Description: Achievement of femoral artery access with AXERA and placement of procedural sheath.
Time Frame: At the time of the femoral artey access procedure up to 1 hour post procedure
Population: Data was not analyzed as the device became unavailable and the study was terminated.
Arm/Group | Standard Manual Compression | AXERA 2 Access System
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Time to Hemostasis
Description: Difference between the time the procedural sheath is removed and hemostasis is observed.
Time Frame: From procedural sheath removal until hemostasis is achieved.
Population: Data not analyzed as the test device became unavailable and the study was terminated.
Arm/Group | Standard Manual Compression | AXERA 2 Access System
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Time to Discharge Eligibility
Description: The time from sheath removal and ambulation to when a subject can be discharged after examination of access site.
Time Frame: Up to 1 day post procedure
Population: Data not analyzed as the test device became unavailable and the study was terminated.
Arm/Group | Standard Manual Compression | AXERA 2 Access System
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Time to Actual Discharge
Description: Time following procedural sheath removal until actual discharge.
Time Frame: Up to 1 day post procedure
Population: Data not analyzed as the test device became unavailable and the study was terminated.
Arm/Group | Standard Manual Compression | AXERA 2 Access System
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Time to Ambulation
Description: Time from sheath removal until the participant can stand or walk 20 feet without rebleeding. Ambulation can be evaluated at 1,2, and 4 hours post sheath removal until the participant can ambulate.
Time Frame: Up to 1 day post procedure
Population: Data not analyzed as the test device became unavailable and the study was terminated.
Arm/Group | Standard Manual Compression | AXERA 2 Access System
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Ability to Sit up at 45-degree Angle
Description: The ability to sit up at a 45-degree angle within 15 minutes of successful hemostasis without rebleed.
Time Frame: 15 minutes of successful hemostasis
Population: Data not analyzed as the test device became unavailable and the study was terminated.
Arm/Group | Standard Manual Compression | AXERA 2 Access System
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Minor Access Site Related Complications
Description: Observation of any minor access site related complications.
Time Frame: Up to 37 days post procedure
Population: Data not analyzed as the test device became unavailable and the study was terminated.
Arm/Group | Standard Manual Compression | AXERA 2 Access System
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Patient Satisfaction
Description: Assessed by a patient satisfaction questionnaire.
Time Frame: Up to 37 days post procedure
Population: Data not analyzed as the test device became unavailable and the study was terminated.
Arm/Group | Standard Manual Compression | AXERA 2 Access System
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Pain Score
Time Frame: Up to 37 days post procedure
Population: Data not analyzed as the test device became unavailable and the study was terminated.
Arm/Group | Standard Manual Compression | AXERA 2 Access System
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Standard Manual Compression | AXERA 2 Access System
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/22
Other Adverse Events (participants affected / at risk) | 1/17 | 2/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Manual Compression (N=17) | AXERA 2 Access System (N=22)
Hematoma (Vascular disorders) | 1 (1) | 1 (1)
Discomfort and paresthesia in groin (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The test device was modified and no longer available to the investigator and the study was terminated. Because of this, secondary outcomes were not analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No